CLINICAL TRIAL: NCT03802851
Title: HoLEP Prior to Radiation Therapy for Patients With LUTS/Retention and Concurrent Prostate Cancer
Acronym: HOLEP-RTPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Bristol Whiles, MD, Principal Investigator, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 143226
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Neoplasms; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: This is a small scale study with initial enrollment of 20 patients in the treatment arm of the study and an additional 10 patients enrolled in the control arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium Laser Enucleation of Prostate (HoLEP) (Experimental): Patients in this arm will undergo holmium laser enucleation of the prostate (HoLEP) for the treatment of lower urinary tract symptoms (LUTS). Patients will undergo HoLEP one time and will return for standard of care follow up.
  Interventions: Procedure: Holmium Laser Enucleation of Prostate (HoLEP)
- Control Arm (No Intervention): Patients in this arm will undergo no additional interventions and will not undergo holmium laser enucleation of the prostate (HoLEP) for the treatment of lower urinary tract symptoms and instead follow standard of care treatment and follow up.

INTERVENTIONS:
Procedure: Holmium Laser Enucleation of Prostate (HoLEP) — Holmium laser enucleation of the prostate (HoLEP) is a surgical treatment use for men with bothersome lower urinary tract symptoms (LUTS) to improve their LUTS. During the procedure a thin telescope-like instrument is inserted into the urethra. The high-powered laser is then inserted through this instrument and used to carefully remove the excess prostate tissue that is causing obstruction of the urethra and contributing to the patient's lower urinary tract symptoms.
  Arms: Holmium Laser Enucleation of Prostate (HoLEP)

SUMMARY:
To determine if holmium laser enucleation of the prostate (HoLEP) for the treatment of lower urinary tract symptoms (LUTS) and/or urinary retention alters the treatment course for patients concurrently diagnosed with prostate cancer.

DETAILED DESCRIPTION:
The investigators propose a prospective trial to investigate pre-radiation holmium laser enucleation (HoLEP) in men with bothersome lower urinary tract symptoms (LUTS) and prostate cancer who have elected for radiation therapy as the primary treatment modality for their prostate cancer. The investigators hypothesize that pre-radiation HoLEP may decrease their overall LUTS and may decrease their need for subsequent radiation therapy. The goal with this study is to better understand the overlap between prostate cancer and LUTS, as well as determine if primary surgical treatment for the LUTS with HoLEP can also serve as a possible treatment modality for concurrent prostate cancer. This information may provide further information to inform future standard of care practices for patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patients must have bothersome lower urinary tract symptoms (LUTS), defined by American Urological Association Symptom Score (AUA SS) of greater than or equal to 15 and/or as defined by a post-void residual of greater than or equal to 350mL and/or as defined by catheter dependence
* Patients must be diagnosed with prostate cancer by pathological tissue analysis
* Patients must have elected for radiation with androgen deprivation therapy as the primary treatment modality for their prostate cancer

Exclusion Criteria:

* Patients who are under 18 years of age are not eligible
* Patients who have a diagnosis of bladder cancer are not eligible.
* Patients with prior treatment for prostate cancer are not eligible.
* Patients with any type of prior prostate surgery (minimally invasive, endoscopic, or otherwise) including prior transurethral resection of the prostate (but excluding prior prostate biopsy) are ineligible.
* Patients with known metastatic prostate cancer are ineligible
* Patients who are enrolled in other surgical or international trials at the time of this study are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Quality of Life - One Year Post Operatively | Quality of life will be assessed one year post-operatively
  The primary object is to determine if holmium laser enucleation of the prostate (HoLEP) improves the quality of life in patients with concurrent prostate cancer who may undergo radiation therapy as well. Quality of life will be assessed using the Expanded Prostate Cancer Index Composite (EPIC) 26. This instrument evaluates patient function and bother after prostate cancer treatment using 26 items and scored on a 0-100 scale, with higher scores indicating a better health related quality of life.
Improvement in Quality of Life - Five Years Post Operatively | Quality of life will be assessed five years post-operatively
  The primary object is to determine if holmium laser enucleation of the prostate (HoLEP) improves the quality of life in patients with concurrent prostate cancer who may undergo radiation therapy as well. Quality of life will be assessed using the Expanded Prostate Cancer Index Composite (EPIC) 26. This instrument evaluates patient function and bother after prostate cancer treatment using 26 items and scored on a 0-100 scale, with higher scores indicating a better health related quality of life.

SECONDARY OUTCOMES:
Prostate Cancer Treatment Course - One Year Post Operatively | Prostate Cancer Treatment Course will assessed one year post-operatively
  The secondary objective is to determine if holmium laser enucleation of the prostate (HoLEP) alters the prostate cancer treatment course in patients. This will assessed by comparing the time from enrollment to the time of initiation of radiation therapy in patients in both arms.
Prostate Cancer Treatment Course - Five Years Post Operatively | Prostate Cancer Treatment Course will assessed five years post-operatively
  The secondary objective is to determine if holmium laser enucleation of the prostate (HoLEP) alters the prostate cancer treatment course in patients. This will assessed by comparing the time from enrollment to the time of initiation of radiation therapy in patients in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Whiles, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States